CLINICAL TRIAL: NCT04935528
Title: Study of Mechanisms of Anti COVID-19 Humoral and Cellular Immune Response Between 1 and 3 Months After Vaccination in a Sample of Patients and Salaried Staff From a French Anti-cancer Center
Brief Title: Mechanisms of Anti COVID-19 Humoral and Cellular Immune Response After Vaccination in a Sample of Patients and Salaried Staff From a French Anti-cancer Center
Acronym: CANSEROVAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-002404-12
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: SARS-CoV-2; vaccination; cellular immune response; humoral response
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vaccined salaried staff (group 1) (Other): vaccined salaried staff group (Distinction between
  * Employees vaccinated with two doses of vaccine (2 Pfizer doses or 2 Astra doses or 1 Pfizer dose + 1 Astra dose) and never infected with SARS-CoV-2
  * And employees vaccinated with one dose of Pfizer or Astra vaccine and previously infected with SARS-CoV-2
  Interventions: Biological: serology and ELISPOT test; Biological: serology
- non vaccined salaried staff (group 2 - witnesses) (Other): non vaccined salaried staff group wtih positive SARS-CoV-2
  Interventions: Biological: serology and ELISPOT test
- vaccined patients (group 3) (Other): vaccined patient group
  Interventions: Biological: serology and ELISPOT test

INTERVENTIONS:
Biological: serology and ELISPOT test — 27 mL blood sample to study the humoral and the cellular immune response
Biological: serology — 7 mL blood sample to study the humoral response
  Arms: vaccined salaried staff (group 1)

SUMMARY:
Special populations are people with a risk to dévelop severe forms of a disease. The immunogenicity and efficacy of vaccines in this population may be different compared of the general population.

For Covid-19, special populations are people with chronic diseases (obesity, diabetes, cancer, etc.) and / or immunocompromised and / or elderly. It is therefore important that the safety of new vaccines as well as their efficacy be evaluated.

Thus, in cancer, most immunosuppressions and immunosuppressive treatments (in particular chemotherapy or certain targeted therapies) risk negatively impacting the effectiveness of the anti-SARS-COV-2 vaccine both for the humoral immune responses (antibodies ) and cellular (T lymphocytes). These patients may develop an insufficient post-vaccination immunity. However, it seems that immunosenescence (ie the aging of the immune system) has little impact on the effectiveness of mRNA vaccines and viral vector vaccines.

The Canserovax study evaluates the impact of anticancer treatments on the quality of the humoral (development of antibodies) and cellular (development of a specific T response) immune response to SARS-CoV-2 in patients treated for cancer after vaccination. It is carried out in patients undergoing treatment and in subjects not suffering from cancer, and not treated for this pathology (vaccinated salaried staff of a french cancer center). The aim is to qualitatively and quantitatively compare the post-vaccination immune responses in these 2 populations.

DETAILED DESCRIPTION:
The main objective of this study is to describe after anti-SARS-CoV-2 vaccination the humoral immune response against the virus (assay of anti-SARS-CoV-2 antibodies to detect the presence and intensity of humoral immune responses) and the cellular response against the virus (specific T response).

Several cohorts are studied:

* Cohort 1 of vaccinated salaried staff (First group : Employees vaccinated with two doses of vaccine (2 Pfizer doses or 2 Astra doses or 1 Pfizer dose + 1 Astra dose) and never infected with SARS-CoV-2) and second group (Employees vaccinated with one dose of Pfizer or Astra vaccine and previously infected with SARS-CoV-2)
* Cohort 2 of unvaccinated salaried staff (controls)
* Cohort 3 of vaccinated cancer patients (metastatic colorectal, metastatic pancreas and metastatic breast cancer)

ELIGIBILITY:
Inclusion Criteria :

Group 1

1. Salaried staff of the Georges-François Leclerc center over 18 years old
2. Subject vaccinated against SARS-CoV-2 for at least 1 month (last injection), AND less than 4 months (last injection).
3. Subject who gave his consent to this study
4. Subject affiliated to a social security scheme

Group 2

1. Salaried staff of the Georges François Leclerc center over 18 years old
2. Subject not vaccinated against SARS-CoV-2
3. Subject having presented a proven infection by SARS-CoV-2 (PCR)
4. Subject who participated in the canSEROcov study with a positive serology result
5. Subject who gave his consent to this study
6. Subject affiliated to a social security scheme

Group 3

1. Patient over 18 years of age treated in Oncology at the GF Leclerc center for:

   * Metastatic colorectal cancer beyond the first line of treatment
   * Metastatic pancreatic cancer as the first line of treatment
   * Metastatic breast cancer treated with anti-CDK4 / 6 + hormone therapy, or localized breast cancer treated with (neo) adjuvant chemotherapy
2. Patient vaccinated against SARS-CoV-2 for at least 1 month (last injection), AND less than 4 months (last injection) with a vaccination performed when the anti-cancer treatment had been started for at least 1 month (last injection) ) (see diagram below)
3. Patient having signed the informed consent for the study
4. Patient affiliated to the social security scheme

Exclusion Criteria:

Groups 1, 2 and 3

1. Minor or under legal protection
2. Person deprived of liberty or under guardianship (including curatorship)
3. Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons (filling in the questionnaire and taking the blood sample)
4. Refusal of the patient or employee to participate
5. pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
seroprevalence of SARS-CoV-2 and ELISPOT | through study completion, an average of 1 year
  rate of specific SARC-Cov-2 IgM and IgG and Human IFN-γ SARS-CoV-2 ELISpot

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges Francois Leclerc, Dijon, France